CLINICAL TRIAL: NCT06185920
Title: Non Interventional Retrospective and Prospective Single Center Descriptive Study of Severe Infections Treated With Phage Therapy at the Hospices Civils de Lyon (PHAGEinLYON Clinic Cohort Study).
Brief Title: PHAGEinLYON Clinic Cohort Study: a Descriptive Study of Severe Infections Treated With Phage Therapy at the HCL.
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0189
Record Dates: First submitted 2023-10-27; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Severe Infection
Keywords: bacteriophage; severe infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe infection.: Patients with severe infection treated with bacteriophage in the Hospices Civils de Lyon from 2015 to 2033.
  Interventions: Other: Description of severe infection

INTERVENTIONS:
Other: Description of severe infection — Description of severe infections treated with bacteriophage in the Hospices Civils de Lyon from 2015 to 2033.

SUMMARY:
PHAGEinLYON Clinic cohort study is a single site non-interventional retrospective and prospective study, initiated by the Hospices Civils de Lyon. Population targeted are patients with a severe infection treated with bacteriophage in the Hospices civils de Lyon from 2015 to 2033. The primary objective is to describe the severe infections treated with phagotherapy. 250 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe infection treated with bacteriophage in the Hospices Civils de Lyon from 01/01/2015 to 01/01/2033
* PHAGEinLYON Clinic cohort study information notice provided to the patient

Exclusion Criteria:

* Opposition of trial participant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 250 patients with severe infection treated with phagotherapy will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2033-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of each type of severe infection | through study completion (5years)
  Rate of each type of severe infection treated with bacteriophage in the Hospices Civils de Lyon from 2015 to 2033.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious and Tropical Diseases of the Croix Rousse Hospital of the Civil Hospitals of Lyon, Lyon, France